CLINICAL TRIAL: NCT00762424
Title: Effect of Tamsulosin on Stone Expulsion and Pain Resolution in ED Patients With Ureterolithiasis
Acronym: Flowmax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WellSpan Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0607030
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Kidney Stone
Keywords: Kidney stone; Ureterolithiasis; Tamsulosin; Flowmax; Emergency Department
MeSH Terms: conditions — Kidney Calculi; Ureterolithiasis; Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tamsulosin (Active Comparator)
  Interventions: Drug: Flowmax
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Flowmax — 0.4 mg once a day until stone passage total = 9 tablets
  Arms: Tamsulosin
Drug: placebo — cornstarch
  Arms: Placebo

SUMMARY:
Tamsulosin (Flowmax)is approved by the FDA for the treatment for enlarged prostate. Several studies regarding the use of Tamsulosin for the treatment of lower kidney stones have been carried out in the non-Emergency Department setting. This study will compare Tamsulosin 0.4 mg with placebo in regards to rate and time of stone passing and will also look at amount of pain. The purpose of this study is to compare the usefulness of Tamsulosin versus placebo on time to stone passage and pain relief in Emergency Department patients with kidney stones.

ELIGIBILITY:
Inclusion Criteria:

* 18 y.o. or older
* diagnosed with a kidney stone less than or equal to 10 mm determined by CT scan
* physician has made the decision that you will be discharged to home
* must be able to take study medication for up to 10 days and strain your urine
* must be able to keep a record of pain medication taken and complete a pain scale rating

Exclusion Criteria:

* patients currently taking: Tamsulosin (Flowmax), calcium channel blockers, beta blockers, alpha blockers, Sildenaphil (Viagara), Tadalaphil (Cilias), Warfarin (Coumadin, Jantoven), Cimetidine (Tagamet, Tagamet HB)
* patients with a clinical and laboratory signs of: urinary tract infection, multiple kidney stones, diabetes, kidney failure, hypotension, pregnancy, fever
* patient known to have hypersensitivity to Tamsulosin
* patient history of cataract surgery
* inability of patient to perform visual pain scale
* allergy or intolerance to acetaminophen/oxycodone
* patient is unable to understand informed consent
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pollack, MD, PhD, Principal Investigator — WellSpan Health
Locations (1):
- York Hospital Emergency Department, York, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tamsulosin | Placebo
Started | 28 | 25
Completed | 28 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: results not available
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamsulosin | Placebo | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Customized [Number; unit: participants]
  >=18 years | 28 | 25 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Time of Stone Passage
Description: Upon discharge, patient must be able to take the medication for 10 days and strain his/her urine. Patient must log the date and time of stone passage, if known.
Time Frame: 10 Days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 28 | 25
hours | 68.8 [0 to 78] | 19.0 [0 to 60]

ADVERSE EVENTS:
Arm/Group | Tamsulosin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/25
Other Adverse Events (participants affected / at risk) | 0/28 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No